CLINICAL TRIAL: NCT02813837
Title: A Multicenter Efficacy and Safety Study of Cluster of Differentiation 19 (CD19)-Targeted CART (CD19CART) Therapy for CD19 Positive Relapsed or Refractory B-cell Hematologic Malignancies (SCT019-01）
Brief Title: Chimeric Antigen Receptor T Cells (CART) Therapy in Refractory/Relapsed B Cell Hematologic Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Innovative Cellular Therapeutics Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCT019-01
Record Dates: First submitted 2016-06-19; First posted 2016-06-27 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Leukemia, B-Cell; Lymphoma, B-Cell
Keywords: relapsed; refractory; CD19+; leukemia; lymphoma
MeSH Terms: conditions — Leukemia, B-Cell; Lymphoma, B-Cell; Recurrence; Leukemia; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- single arm (Experimental): Experimental: CD19 CART cell.The target dose range administered in this study is 1x10e5-1x10e7 CART-19 cells/kg.
  Interventions: Biological: CD19CART

INTERVENTIONS:
Biological: CD19CART — Patients will be given infusions of CD19CART cells into the vein over a period of 1 to 3 days. The target dose range administered in this study is 1x10e5-1x10e7 CD19CART cells/kg. Patients will be monitored for a response, toxic effects, and the expansion and persistence of circulating CD19CART cells.
  Other Names: CD19-directed chimeric antigen receptor modified T cells

SUMMARY:
This single arm, open-label, multi-center clinical trial is studying CD19 targeted chimeric antigen receptor T cells therapy in treating patients with CD19 positive malignant B-cell derived leukemia and lymphoma that is relapsed (after stem cell transplantation or chemotherapy) or refractory to chemotherapy.

DETAILED DESCRIPTION:
This single arm, open-label, multi-center clinical trial is studying CD19 targeted chimeric antigen receptor T cells therapy in treating patients with CD19 positive malignant B-cell derived leukemia and lymphoma that is relapsed (after stem cell transplantation or chemotherapy) or refractory to chemotherapy. When patients enroll in this trial, autologous CD19CART cells were generated from the mononuclear cells of the patient's peripheral blood (PB). During the term of cell preparation of CD19CART cells, patients will receive a conditioning regimen. One day after completing conditioning regimen, the patient will be given infusions of CD19CART cells into the vein over a period of 1 to 3 days. Patients will be monitored for a response, toxic effects, and the expansion and persistence of circulating CD19CART cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as CD19 positive refractory and relapsed B cell hematologic malignancies included acute lymphoblastic leukemia (ALL),chronic lymphocytic leukemia(CLL),non-Hodgkin's lymphoma(NHL)
* not eligible or appropriate for auto-HSCT or allo-HSCT or relapsed after hematopoietic stem cell transplant(HSCT)
* At least one measurable lesion defined as one lesion larger than 1.5cm or two lesion more than 1.0cm(for patients with NHL )
* Age ≤60 years
* Eastern Cooperative Oncology Group(ECOG) Performance status 0 to 2, Expected survival > 6 months
* Left Ventricular Ejection Fraction (LVEF) > 50%
* no history of other malignancies;
* no other serious diseases which conflict with the treatment in the present trial
* All patients should consent to adopt efficient contraception methods during the treatment and after the treatment. The pregnant tests of women who are in child bearing period should be negative before the treatment.
* patients should understand and are willing to participate in the trial. Inform consent form is supposed to obtained before treatment

Exclusion Criteria:

* Diagnosis or classification undefined
* Those with primary central nervous system lymphoma or testicular leukaemia or lymphoma
* Patients with a known history or prior diagnosis of epilepsia or other disease affecting the central nervous system, or serious mental diseases;
* Patients who have secondary leukaemia or lymphoma after chemotherapy or radiotherapy for other malignancies
* Active acute or chronic graft-versus-host disease (GVHD) requiring systemic therapy, concurrent use of immunosuppressant medications
* Class III/IV cardiovascular disability according to the New York Heart Association Classification
* Pregnant or lactating women(the safety of this therapy on unborn children is not known)
* With active infection
* Active hepatitis B, hepatitis C or syphilis infection
* Patients use of systemic steroids within 2 weeks. Recent or current use of inhaled steroids is not exclusionary
* Prior treatment with gene therapy product
* Cluster of differentiation 3(CD3) positive cells<0.9x10^4/ml in peripheral blood (PB)
* Organ function meeting following criteria: liver and renal function: alanine aminotransferase(ALT)/aspartate aminotransferase(AST) > 3 times the upper limit of normal, or bilirubin>2.0 mg/dl（34.2umol/L）, or creatinine >2.5mg/dl（221.0umol/L） ; hematopoietic function:Neutrophil count<1.0x10^9/L，hemoglobin<80g/L，platelet <50x10^9/L(for patients with NHL )
* Any uncontrolled active medical disorder that would preclude participation as outlined
* HIV infection
* The researchers considered unsuitable to participate in this clinical study.
* Patients with poor compliance

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-06; Primary Completion 2021-01 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | up to 12 months

SECONDARY OUTCOMES:
Anti-leukemia or lymphoma responses to CD19CART cell infusions | up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hu, Ph.D, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; He Huang, Ph.D, Study Director — The First Affiliated Hospital of the College of Medicine, Zhejiang University
Locations (1):
- Innovative Cellular Therapeutics CO., LTD., Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided